CLINICAL TRIAL: NCT05935501
Title: Safety and Efficacy of Formaderm Young Dermal Filler Injection for the Correction of Moderate-to-severe Facial Wrinkles.
Brief Title: Clinical Trial of Cross-linked Hyaluronic Acid Dermal Filler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maxigen Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBI-2016-01
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Hyaluronic Acid; Dermal Fillers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Formaderm Young (Experimental): Formaderm Young was randomly administered to subjects. The injection volume was limited to 2c.c.
  Interventions: Device: Formaderm Young
- Restylane (Active Comparator): Restylane was randomly administered to subjects. The injection volume was limited to 2c.c.
  Interventions: Device: Restylane

INTERVENTIONS:
Device: Formaderm Young — Dermal filler injection to facial areas.
  Arms: Formaderm Young
Device: Restylane — Dermal filler injection to facial areas.
  Arms: Restylane

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of Formaderm Young Dermal Filler Injection, which is a hyaluronic acid dermal filler injected into the mid to deep dermis for the correction of moderate-to-severe nasolabial fold facial wrinkles.

The main questions it aims to answer are:

* The differences of Wrinkle Severity Rating Scale (WSRS) after the injection.
* The treatment improvement assessed by Global Aesthetic Improvement Scale (GAIS).
* Safety Indicators of which incidences on the day of the injection or after the injection.

Participants will be blinded and randomized into either experiment group or control group, and re-visited on 1, 3, 6, 9 and 12 month after injection.

Researchers will compare if the test product is non-inferiority to Restylane.

DETAILED DESCRIPTION:
A prospective, parallel, two-center, non-inferior, randomized, double-blind trial was conducted in this study. It was planned to recruit 157 subjects for each group, considering a 10% dropout rate that would lead to 320 subjects overall.

Subjects eligible in the screening will be enrolled. Each patient will receive the same treatment, either Formaderm Young Dermal Filler Injection or Restylane, to correct both sides of the nasolabial fold through randomization.

Clinical efficacy will be assessed by the blinded physician using the WSRS and GAIS, as well as by subjects using GAIS. The safety issue of Formaderm Young or Restylane will be identified and recorded during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are aged 18-65 years old of both sexes.
* Subjects who are willing to undergo both sides nasolabial fold therapy.
* The baseline measurement on the wrinkle severity rating scale (WSRS) should be 3-4 points, and the left and right sides should exhibit symmetry.
* Willing to comply with re-visit schedule and sign the informed consent.

Exclusion Criteria:

* Women subjects who are pregnant, breastfeeding, planning to become pregnant, and not willing to take contraception during the trial period.
* Those who are emotionally unstable or suffering from a mental disease.
* Those who have unhealthy facial skin or severe skin disease, inflammation, or related symptoms such as infections, psoriasis, herpes, and similar conditions.
* Those with any disease that would interfere the assessment of skin aging.
* Those who have a scar in the nasolabial fold area.
* Those with connective tissue diseases.
* Those with diabetes or systemic disease that cannot be controlled.
* Those suffering from immunity related disorder.
* Those with a scar-prone constitution.
* Patients undergoing anticoagulant treatment, those who have a medical history of coagulation defects.
* Patients taking antiplatelet medicine that could affect platelet function, such as Aspirin or non-steroidal anti-inflammatory analgesics.
* Those with a allergy history of cosmetic filling agent, any type of hyaluronic acid implants or local anesthetic.
* Those who have undergone facial cosmetic treatments or surgery before the trial:
* Chemical or physical treatments that affect local configuration before the trial, such as laser procedures, skin resurfacing, chemical peel or Face Wrinkle Correction Surgery within 6 month.
* Facial surgery or dermal filler at nasolabial fold area within 12 month.
* Those who have cosmetic surgery with silicone in their body or material that cannot be absorbed by the body (permanent filling agent).
* Those who are not willing to avoid undergoing other cosmetic treatment and surgery, such as facial filling, botulinum toxin Injection, laser procedures, chemical peel or facelift surgery.
* Those who have participate in another clinical investigation within 12 month.
* Those who are deemed unfit for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
WSRS improvement ratio at 6 month post-injection | Baseline and 6 month post-injection
  The difference of WSRS(Wrinkle Severity Rating Scales) between baseline and 6 month post-injection. A positive value indicated"effective" improvement; while a value of 0 or a negative value was regarded as "ineffective" treatment. And the WSRS improvement ratio was defined as the effective improvement ratio of either group.

SECONDARY OUTCOMES:
WSRS score | Baseline and 1 month, 3month, 6month post-injection
  Blinded physician rated the score of WSRS(Wrinkle Severity Rating Scales) for both group respectively. The WSRS is a 5-grade instrument for facial wrinkle, Grade 1(absent, no visible nasolabial fold; continuous skin line ) to Grade 5(extreme, extremely deep and long nasolabial fold, detrimental to facial appearance;2-4mm visible V-shaped fold when stretched; unlikely to have satisfactory correction with injectable implant alone).
WSRS improvement ratio | Baseline, 1 month and 3month post-injection
  The difference of WSRS(Wrinkle Severity Rating Scales) between baseline and 1 month and 3 month post-injection. A positive value indicated "effective" improvement; while a value of 0 or a negative value was regarded as "ineffective" treatment. And the WSRS improvement ratio was defined as the effective improvement ratio of either group.
GAIS score assessed by physician | Baseline, 1 month, 3month and 6month post-injection
  Compared with the baseline photographs, blinded physician rated the class of GAIS(Global Aesthetic Improvement Scale) from 5(exceptional improvement, excellent corrective result) to 1(worsened patient, the appearance has worsened compared with the original condition) for both group at 1 month, 3 month and 6 month post-injection respectively.
GAIS score assessed by subjects | Baseline, 1 month, 3month and 6month post-injection
  Compared with baseline, subjects themselves rated the class of GAIS(Global Aesthetic Improvement Scale) from 5(exceptional improvement, excellent corrective result) to 1(worsened patient, the appearance has worsened compared with the original condition) for both group at 1 month, 3 month and 6 month post-injection respectively.
Incidence of Treatment-related Adverse Events | Month 0 to month 12
  The adverse events are defined as any unfavorable sign occurrence in a subject after treatment. The investigator assesses the severity and the relationship of each event to the use of the study device.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Chaoyang
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Tongren